CLINICAL TRIAL: NCT02061501
Title: Evaluation of the Efficacy of Optometric Rehabilitation on Visual Cognitive Deficits in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5542
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Visual Cognitive Deficits
Keywords: visual cognitive deficits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Speech therapy (Active Comparator): Speech therapy (30 min per week) alone for the 6 first months. Then speech therapy (30 min per week) and optometric therapy (30 min per week) for the 6 last months.
  Interventions: Other: Optometric therapy during 6 months
- Speech therapy and optometric therapy (Experimental): Speech therapy (30 min per week) and optometric therapy (30 min per week) for 12 months.
  Interventions: Other: Optometric therapy during 12 months

INTERVENTIONS:
Other: Optometric therapy during 6 months — Optometric therapy during 6 months, once a week
  Arms: Speech therapy
Other: Optometric therapy during 12 months — Optometric therapy once a week, during 12 months
  Arms: Speech therapy and optometric therapy

SUMMARY:
Visual cognitive deficits in children are frequent, with an impact on working and daily activities. Optometric therapy may improve those functions, however few studies have been performed.

We aim to evaluate the efficacy of such therapy by a comparative study between two groups of children aged between 5 and 12 after 6 months of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* visual cognitive deficits
* normal intelligence

Exclusion Criteria:

* cerebral palsy
* mental deficiency
* visual acuity deficit

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Calculation of a composite score at Visit 1 | Visit 1 (6 months of rehabilitation)
  The composite score is calculated from the results obtained at several neuropsychology and optometric tests.
  Basal score is calculated at Visit 0 (inclusion visit).

SECONDARY OUTCOMES:
Calculation of a composite score at Visit 2 | Visit 2 (12 months of rehabilitation)
  The composite score is calculated from the results obtained at several neuropsychology and optometric tests.

OTHER OUTCOMES:
Quality of life | Visit 2 (12 months of rehabilitation)
  Quality of life assessed by a questionnaire at V0, V1 and V2.

CONTACTS AND LOCATIONS:
Locations (1):
- CRTLA - Hôpital de Hautepierre- CHRU Strasbourg, Strasbourg, France